CLINICAL TRIAL: NCT05987735
Title: BLAME-LESS STUDY: a Two-arm Randomized Controlled Trial Evaluating the Effects of an Online Psycho-education Program for Adolescents Who Experienced (sexual) Violence.
Brief Title: Psycho-education Program BLAME-LESS and It's Effect on Traumarelated Shame and Guilt
Acronym: BLAME-LESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ontschuldig
Record Dates: First submitted 2023-07-05; First posted 2023-08-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Trauma
Keywords: Shame; Guilt; Defense Response; Defense Cascade; PTSD; Psycho-education; Tonic Immobility; Appeasement
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: a two-arm randomized controlled trial (RCT). . Participants will be randomized into either the intervention group or waiting-list control group. If allocated to the intervention group, participants will have direct access to the online intervention for two weeks after allocation. When a participant is assigned to the waiting-list control group, he or she has a two-week waiting period, after which the participant will have access to the intervention. Assessments take place after screening (T0), at baseline (T1), and two weeks after allocation (T2). Participants in the waiting-list group will also be assessed two weeks after they have gained access to the intervention (T3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLAME-LESS Program (Experimental): If allocated to the intervention group, participants will have direct access to the online intervention for two weeks after allocation.
  Interventions: Behavioral: BLAME-LESS
- Waiting-list control group (No Intervention): When a participant is assigned to the waiting-list control group, he or she has a two-week waiting period, after which the participant will have access to the intervention.

INTERVENTIONS:
Behavioral: BLAME-LESS — The BLAME-LESS program was designed to educate about common defense responses that may occur during and after (sexual) violence. The main goal of the program is to reduce the feelings of shame and/or guilt related to these responses. The program was created in collaboration with licensed developmental and clinical psychologists with extensive psycho-trauma expertise, young adults who are experienced experts, visual artists, and web designers. The program is offered via a website and consists of three modules.
  Arms: BLAME-LESS Program

SUMMARY:
The primary objective of the BLAME-LESS study is to examine the effectiveness of an online psychoeducation program in reducing trauma-related feelings of shame and guilt in adolescents who experienced sexual or physical abuse .

DETAILED DESCRIPTION:
The study follows a two-arm RCT (n=34). The effects of a brief online psychoeducation program will be compared, with a waiting-list control group. The intervention aims to reduce feelings of trauma-related shame and guilt that adolescents experience regarding their own defense responses during and after (sexual) violence. Assessments take place after screening, at baseline, two weeks after allocation to the intervention or waiting-list, and, only for the waiting-list participants, seven weeks after allocation to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* the participant experienced one or more traumatic life events, including (sexual) violence as indicated by the CTSQ;
* the participant reported one or more feelings of guilt and/or shame on the CERQ (items 1 and/or 10 and/or 19 and/or 28)
* the participant being fluent in written and spoken Dutch;
* the participant is motivated and available for a period of seven weeks to engage in the study, including the psychoeducation program BLAME-LESS, and commit to the assessments.

Exclusion Criteria:

* acute suicidal behavior or suicidal ideations requiring immediate hospitalization;
* the participant has already read the book that this program is based upon: "Paralyzed with Fear" (In Dutch: Verlamd van Angst, van Minnen 2017), or has been intensively informed otherwise in the past 12 months by a psychologist about common defense responses during and after trauma;
* Cognitive Impairments (IQ < 70);
* the participant has a brother or sister in the present study;
* the participant is already involved in trauma-focused treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Changes in Feelings of Shame and Guilt | The SGATS will be assessed at before treatment (T1 = Week 1), after treatment (T2 = Week 4, T3 = week 7)
  The primary objective of the BLAME-LESS study is to examine the effectiveness of an online psychoeducation program, BLAME-LESS, compared to a waiting-list control group of adolescents (12 - 18 years) who experienced sexual or physical abuse in reducing trauma-related feelings of shame and guilt. The Shame and Guilt After Trauma Scale (SGATS) (Aakvaag et al., 2016) measures trauma-related shame and guilt. The SGATS consists of nine items, four on trauma-related feelings of shame and five on trauma-related feelings of guilt (Aakvaag et al., 2016). Each question can be answered on a 3-point Likert scale (0 = no, 1 = yes, a little, 2 = yes, a lot).

SECONDARY OUTCOMES:
Secondary outcome: Changes in Posttraumatic Stress Symptoms | The KJTS will be assessed before treatment (T1 = Week 1) and after treatment (T2 = Week 4, T3 = Week 7).
  The second objective of the research is to examine the effects of the intervention on PTSD symptoms. The Dutch version of the Child and Adolescent Trauma Screener (KJTS-NL; Kooij & Lindauer, 2019) is a questionnaire for children and adolescents that serves as a screening tool for PTSD symptoms (Sachser et al., 2017). The severity of PTSD symptoms is measured with 20 items, rated on a 4-point Likert scale (range 1-4). A total score below 15 suggests no (clinical) indication of the presence of a PTSD classification, a score between 15 and 20 suggests the possible presence of a clinical PTSD classification, and a score above 20 suggests an increased chance of the presence of a PTSD classification.
Secondary outcome: Changes in Depression and Anxiety Symptoms | The PROMIS will be assessed before treatment (T1 = Week 1) and after treatment (T2 = Week 4, T3 = Week 7)
  The third objective of the research is to examine the effects of the intervention on anxiety and depression symptoms. The Patient-Reported Outcomes Measurement Information System (PROMIS; Terwee et al., 2014) measures Anxiety and Depression symptoms. The lists consist of a dynamic set of item banks based on Computerized Adaptive Testing (CAT). Both questionnaires consist of 8 items. Each question can be answered as follows: never, almost never, sometimes, often, very often.
Secondary outcome: Changes in Posttraumatic Cognition | The CPTCI will be assessed before treatment (T1 = Week 1) and after treatment (T2 = Week 4, T3 = Week 7)
  The fourth objective of the research is to examing the effects of the intervention on posttraumatic cognitions. The Child Posttraumatic Cognitions Inventory (CPTCI; Meiser-Stedman et al., 2009) is a self-report questionnaire that measures trauma-related cognitions in children and adolescents. The questionnaire consists of two subscales (permanent and disturbing change subscale, CPTCI-PC; fragile person in a scary world subscale, CPTCI-SW) with a total of 25 items that can be answered on a four-point Likert scale (ranging from 1 (strongly disagree) to 4 (strongly agree). The English version of the CPTCI has been validated in children aged-6-18 years. The Dutch CPTCI has good reliability and validity (Diehle et al., 2015), high internal consistency (Cronbach's alpha 0.86-0.93), and good convergent validity.
Secondary outcome: Changes in motivation and disclosure | The TPEQ will be assessed before treatment (T1 = Week 1) and after treatment (T2 = Week 4, T3 = Week 7)
  The fifth objective of the research is to examing the effects of the intervention on motivation to engage in traumafocused treatment and to disclose traumatic memories. The Treatment Program and Evaluation Questionnaire (TPEQ; Murphy et al., 2009) assesses readiness and motivation for trauma-focused treatments (Murphy et al., 2009). The questions were answered on a 7-point Likert scale (ranging from 1 = strongly disagree to 7 = strongly agree). A higher score indicates greater willingness and motivation for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nanda Lambregts-Rommelse, Prof.dr, Principal Investigator — Karakter Kinder- en Jeugdpsychiatrie
Locations (1):
- Karakter kinder- en jeugdpsychiatrie, Almelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No